

# STATISTICAL AND EPIDEMIOLOGICAL ANALYSIS PLAN (SEAP) FOR NON-INTERVENTIONAL STUDIES (NIS)

| <u> </u> | |
|---|---|
| Document Number: | c40729787-01 |
| BI Study Number: | 1237-0110 |
| BI Investigational<br>Product(s) | Spiolto Respimat |
| Title: | Effectiveness of Maintenance Treatment with Tiotropium + Olodaterol in Comparison to Inhaled Corticosteroids + Longacting β2 agonists in COPD patients in Taiwan: a non-interventional study based on the Taiwan National Health Insurance (NHI) data. |
| Brief lay title: | Effectiveness of Tiotropium + Olodaterol versus ICS+LABA among COPD patients in Taiwan. |
| SEAP version identifier: | 1.0 |
| Date of last version of SEAP: | Not applicable |
| NIS Statistician [SEAP author] | The SEAP is prepared by the principal investigator, an epidemiologist, but not a statistician. |
| NIS Lead<br>[SEAP reviewer] | |
| NIS Data Manager<br>[SEAP reviewer] | |


Proprietary confidential information

© 2022 Boehringer Ingelheim Group of companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### **TABLE OF CONTENTS**

| TITL | E PAGE1 |
|---|---|
| TABI | LE OF CONTENTS |
| 1. | LIST OF ABBREVIATIONS |
| 2. | RESPONSIBLE PARTIES |
| 3. | PURPOSE AND SCOPE |
| 4. | AMENDMENTS AND UPDATES 4 |
| 5. | RESEARCH QUESTION AND OBJECTIVE4 |
| 6. | RESERACH METHODS4 |
| 6.1 | STUDY DESIGN4 |
| 6.2 | SETTING5 |
| 6.3 | STUDY POPULATION5 |
| 6.4 | STUDY VISITS8 |
| 7. | VARIABLES8 |
| 7.1 | EXPOSURES8 |
| 7.2 | OUTCOMES8 |
| 7 | .2.1 Primary outcomes |
| 7 | .2.2 Secondary outcomes |
| 7.3 | COVARIATES |
| 7.3<br>8. | COVARIATES 11 DATA SOURCES 13 |
| 7.3<br>8.<br>9. | COVARIATES |
| 7.3<br>8.<br>9. | COVARIATES |
| 7.3<br>8.<br>9.<br>9.1<br>9.2 | COVARIATES |
| 7.3<br>8.<br>9.<br>9.1<br>9.2<br>9.3 | COVARIATES |
| 7.3<br>8.<br>9.<br>9.1<br>9.2<br>9.3 | COVARIATES |
| 7.3<br>8.<br>9.<br>9.1<br>9.2<br>9.3 | COVARIATES |
| 7.3<br>8.<br>9.<br>9.1<br>9.2<br>9.3<br>10. | COVARIATES |
| 7.3<br>8.<br>9.<br>9.1<br>9.2<br>9.3<br>10.<br>10.1 | COVARIATES |
| 7.3<br>8.<br>9.<br>9.1<br>9.2<br>9.3<br>10.<br>10.1 | COVARIATES |
| 7.3<br>8.<br>9.<br>9.1<br>9.2<br>9.3<br>10.<br>10.1 | COVARIATES |
| 7.3<br>8.<br>9.<br>9.1<br>9.2<br>9.3<br>10.<br>10.1<br>10.3<br>11.<br>12. | COVARIATES 11 DATA SOURCES 13 DATA MANAGEMENT AND SOFTWARE/TOOLS 14 SOFTWARE/TOOLS 14 HANDLING OF MISSING VALUES 14 HANDLING OF INCONSISTENCIES IN DATA AND OUTLIERS 14 DATA ANALYSIS 14 MAIN ANALYSIS 14 SAFETY ANALYSIS 21 QUALITY CONTROL 21 REFERENCES 21 PUBLISHED REFERENCES 21 |
| 7.3<br>8.<br>9.<br>9.1<br>9.2<br>9.3<br>10.<br>10.1<br>11.<br>12.<br>12.1<br>12.2 | COVARIATES 11 DATA SOURCES 13 DATA MANAGEMENT AND SOFTWARE/TOOLS 14 SOFTWARE/TOOLS 14 HANDLING OF MISSING VALUES 14 HANDLING OF INCONSISTENCIES IN DATA AND OUTLIERS 14 DATA ANALYSIS 14 MAIN ANALYSIS 14 SAFETY ANALYSIS 21 QUALITY CONTROL 21 REFERENCES 21 PUBLISHED REFERENCES 21 UNPUBLISHED REFERENCES 22 |
| 7.3<br>8.<br>9.<br>9.1<br>9.2<br>9.3<br>10.<br>10.1<br>11.<br>12.<br>12.1<br>12.2<br>ANN | COVARIATES 11 DATA SOURCES 13 DATA MANAGEMENT AND SOFTWARE/TOOLS 14 SOFTWARE/TOOLS 14 HANDLING OF MISSING VALUES 14 HANDLING OF INCONSISTENCIES IN DATA AND OUTLIERS 14 DATA ANALYSIS 14 MAIN ANALYSIS 14 SAFETY ANALYSIS 21 QUALITY CONTROL 21 REFERENCES 21 PUBLISHED REFERENCES 21 |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 1. LIST OF ABBREVIATIONS

BI Boehringer Ingelheim CI Confidence Interval

COPD Chronic Obstructive Pulmonary Disease
DMRP Data management and review plan

ICS Inhaled corticolsteroids
IQR Interquartile range
LABA Long-acting β2-agonists

LAMA Long-acting muscarinic antagonists
NHI Taiwan National Health Insurance

NIS Non-interventional study

Olo Olodaterol

PS Propensity score

SEAP Statistical and epidemiological analysis plan

Tio Tiotropium

#### 2. RESPONSIBLE PARTIES

| NIS Statistician [SEAP author]: | | the principal | investigator | who | is an |
|---|---|---|---|---|---|
| epidemiologist and not a statisticia | n | | | | |

#### SEAP reviewers are:

- BI NIS Lead [SEAP reviewer] (in all cases):
- NIS Data Manager [SEAP reviewer] (in all cases):
- RWE CoE [SEAP reviewer] (for all globally initiated studies and for local studies) involving BI products and Global NIS not involving BI products:
- TSTAT (for NISnd only):NA
- TM Epi [SEAP reviewer] (When BI NIS lead is not TM Epi; in all cases):

#### 3. PURPOSE AND SCOPE

COPD is a leading cause of morbidity and mortality throughout the world. The role of ICS in COPD has been debated for decades and studies have been conducted to investigate the effect

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

of ICS-containing therapy in patients with COPD. The aim of this real world study is to assess effectiveness and safety profile between inhaled tiotropium/olodaterol (Tio/Olo) and corticolsteroids / long-acting  $\beta$ 2-agonists (CS/LABA).

#### 4. AMENDMENTS AND UPDATES

None

## 5. RESEARCH QUESTION AND OBJECTIVE

#### **Primary objective:**

 To compare time to the first moderate or severe COPD exacerbations between initiators of Tio/Olo and ICS/LABA after entry between 1<sup>st</sup> January 2014 and 31<sup>st</sup> December 2019

#### **Secondary objectives:**

- To compare time to escalation to triple therapy between initiators of Tio/Olo and ICS/LABA;
- To compare the rate of escalation to triple therapy between initiators of Tio/Olo and ICS/LABA;
- To compare the time to first hospitalization for community-acquired pneumonia between initiators of Tio/Olo and ICS/LABA;
- To compare the number of prescriptions of rescue medication between initiators of Tio/Olo and ICS/LABA
- To compare the annualized rate of moderate or severe COPD exacerbation

The study period between 1<sup>st</sup> January 2014 and 31<sup>st</sup> December 2019 apply to secondary objectives above.

#### 6. RESEARCH METHODS

#### 6.1 STUDY DESIGN

This study will be a non-interventional cohort study using Taiwan National Health Insurance (NHI) claims database, Taiwan Cancer Registry (TCR) and Taiwan Mortality Data. It is a secondary health data environment with relevant information on treatment and disease outcomes of COPD patients among a population of predominantly ethnic Han Chinese. As a publicly funded single payor health insurance program, a wide range health services, including hospital care, emergency visits, ambulatory clinic services, and prescription drugs are covered for virtually all Taiwan residents. The complete capture of health care encounters reimbursed by NHI among a defined group of patients has served as the basis of many longitudinal studies that evaluated safety profiles of prescribed medications.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Health data that are available for research are provided by the Health and Welfare Data Science Center (HWDSC) of the Department of Statistics, Ministry of Health and Welfare. The HWDSC staff encrypt the national ID for all individuals according to a secure encryption algorithm that is specific for each study, and the encrypted ID all individuals is used for linkage between databases. While the study will provide safety data on drugs of interest, from a regulatory perspective the source data are not auditable, nor de-identified individual level data be brought outside of HWDSC for independent verification of analysis.

Limitations of health insurance databases are well-known, as there is no information on results of clinical parameters (such as blood pressure and body mass index), clinical examinations (such as spirometry findings), or life style attributes (such as smoking). A specific items that needs to be considered for this particular study project is whether the findings are generalizable to COPD patients in China. While there is high similarity between COPD patients in Taiwan and those in China in terms of ethnicity and dietary patterns, management patterns for COPD patients, including comorbid conditions, concomitant medications, and use of traditional Chinese medication regimens, may be different.

Taking into account the strengths and potential limitations of the data source, the population-based nature and potentially large study size of patients on drugs of interest are the major reasons that this data source is a viable option for the study.

#### 6.2 SETTING

Incident Tio/Olo combined inhaler or a ICS/LABA combined inhaler use would be identified from the Taiwan National Health Insurance (NHI) claims data through 2014 to 2019, with a 1-year look-back period to define new user.

#### 6.3 STUDY POPULATION

#### **Inclusion Criteria:**

- 1. At least one prescription for Tio/Olo combined inhaler or a LABA/ICS combined inhaler between 1st January 2014 and 31st December 2019.
  - a) The first dispensing of either Tio/Olo or LABA/ICS combined inhaler will be defined as the index date;
  - b) For the main analyses, only fixed dose combination (FDC) inhalers will be included.
- 2. Aged  $\geq$  40 years on the index date
- 3. At least one diagnosis of COPD (ICD9: 491.x, 492.x, 496; ICD10: J41.x, J42, J43.x, J44.x) at any time prior to or on the index date;

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 4. At least one year of continuous medical and health insurance plan prior to the index date will be required to allow for a look-back period for the covariates and identification of new use of the study drugs;
- 5. At least one record in the health insurance system database.

#### **Exclusion Criteria:**

- 1. Any use of LAMA/LABA, ICS/LABA, or ICS/LAMA/LABA in free or fixed form for one year prior to the index date (the free combination will be defined as the prescriptions of the interest products within 30 days of each other);
- 2. Individuals with asthma, allergic rhinitis, lung cancer, interstitial lung disease, or lung transplant identified at any time prior to the index date

Relevant ICD codes and procedure code are provided in the Annex.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c40729787-01 

Figure 1. Patient selection flow chart



Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 6.4 STUDY VISITS

Not applicable.

#### 7. VARIABLES

#### 7.1 EXPOSURES

Exposure of this study is defined as new initiation of Tio/Olo or ICS/LABA (FDC) during the study period. Detailed drug codes are provided in the Annex.

#### 7.2 OUTCOMES

#### 7.2.1 Primary outcomes

#### > Time to the first moderate or severe COPD exacerbations after index date

The definition of moderate or severe COPD exacerbation:

- a. Moderate exacerbations will be defined as an outpatient visit with a diagnosis code for COPD in any field + a prescription for an oral corticosteroid or an antibiotic for respiratory infections
- b. Severe exacerbations will be defined as a hospitalization or emergency room visit with a primary diagnosis for COPD

Detailed diagnosis codes are listed in Annex.

Tio/Olo users will be matched to the comparator through 1:1 propensity score matchingFor the analysis of the primary outcome, individuals will be followed up from the index date until the first moderate or severe COPD exacerbation. For detailed, please refer to section 10.1. As time-to-event data, the main analysis will be univariate proportional hazard regression analysis to estimate the hazard ratio (Tio/Olo vs. comparator) and its 95% confidence interval (CI). Detailed analytic approach is described in Section 10.1.

### 7.2.2 Secondary outcomes

### Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Analysis of the secondary outcomes will be applied to the propensity-score matched cohorts developed for the primary outcome of interest. Detailed description of the analysis approach is described in Section 10.1

#### (1). Time to triple therapy escalation after index date

Triple therapy escalation, defined as any LAMA/LABA/ICS fixed dose combination or any concurrent use for 30 consecutive days of the following:

- a. any LAMA/LABA fixed dose combination + any ICS single formulation
- b. any LAMA single formulation + any LABA/ICS fixed dose combination
- c. any LAMA single formulation + any LABA single formulation + any ICS single formulation

The event date will be the 30<sup>th</sup> day after initiation of triple therapy.

As time-to-event data, the analysis will be univariate proportional hazard regression analysis to estimate the hazard ratio (Tio/Olo vs. comparator) and its 95% CI.

#### (2). Incidence rate of triple therapy initiation (first event per patient)

Triple therapy escalation, defined as any LAMA/LABA/ICS fixed dose combination or any concurrent use for 30 consecutive days of the following:

- a. any LAMA/LABA fixed dose combination + any ICS single formulation
- b. any LAMA single formulation + any LABA/ICS fixed dose combination
- c. any LAMA single formulation + any LABA single formulation + any ICS single formulation

For incidence rates, it will be calculated for each cohort as follows:

Incidence rate among the Tio+Olo cohort = (total number of patients in the Tio+Olo cohort experiencing an event of interest for the first time during the given time period) / (total person-time at risk from current use of Tio+Olo during the given period)

Incidence rate among the comparison cohort = (total number of patients in the comparator LABA/ICS cohort experiencing an event of interest for the first time during the given time period) / (total person-time at risk from current use of comparator LABA/ICS during the given period)

The incidence rate ratio (IRR) and incidence difference for the outcome in the Tio+Olo - exposed group relative to that in the comparator group will be derived as follows:

Incidence rate ratio = incidence rate from the Tio+Olo cohort divided by the incidence rate from the matched comparator cohort.

Incidence difference = incidence rate from the Tio+Olo cohort – incidence rate from the matched comparator cohort

### Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The IRR and their 95% CIs will be calculated using univariate negative binomial model. Incidence differences and their 95% confidence intervals will also be derived.

#### (3). Time to first hospitalization for community-acquired pneumonia after entry

Community-acquired pneumonia related diagnosis codes and operational definition are listed in the Annex.

As time-to-event data, the analysis will be univariate proportional hazard regression analysis to estimate the hazard ratio (Tio/Olo vs. comparator) and its 95% confidence interval (CI).

#### (4). Annualized rate of prescriptions of rescue medications after the index date

Rescue medications are defined as free or combination use of SABA or SAMA. Detailed drug ATC codes are listed in Annex.

For annualized rates, it will be calculated for each cohort as follows:

Annualized rate among the Tio+Olo cohort = (total number of events in the Tio+Olo cohort during the given time period) / (total person-year at risk from current use of Tio+Olo during the given period)

Annualized rate among the comparison cohort = (total number of events in the comparator LABA/ICS cohort during the given time period) / (total person-year at risk from current use of comparator LABA/ICS during the given period)

For annualized rate and total number of prescriptions of rescue medications, the rate ratio of Tio+Olo – exposed group relative to LABA/ICS group, along with 95% CI will be derived using univariate negative binomial model.

#### (5). Annualized rate of moderate or severe COPD exacerbation after the index date

The definition of moderate or severe COPD exacerbation:

- a. Moderate exacerbations will be defined as an outpatient visit with a diagnosis code for COPD in any field + a prescription for an oral corticosteroid or an antibiotic for respiratory infections, prescriptions within 30 days of each other were considered as continuation of the initial exacerbation.
- b. Severe exacerbations will be defined as a hospitalization or emergency room visit with a primary diagnosis for COPD; hospitalizations or emergency room visits within 30 days of each other were considered as continuation of the initial exacerbation.

For annualized rates, it will be calculated for each cohort as follows:

Annualized rate among the Tio+Olo cohort = (total number of events in the Tio+Olo cohort during the given time period) / (total person-year at risk from current use of Tio+Olo during the given period)

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Annualized rate among the comparison cohort = (total number of events in the comparator LABA/ICS cohort during the given time period) / (total person-year at risk from current use of comparator LABA/ICS during the given period)

For annualized rate of moderate or severe COPD exacerbations, the rate ratio of Tio+Olo – exposed group relative to LABA/ICS group, along with 95% CI will be derived using negative binomial model.



#### 7.3 COVARIATES

Demographic characteristics and cohort entry information:

- Sex
- Age
- Calendar year of cohort entry
- Season of index date (winter, Dec-Feb; spring, Mar-May; summer, Jun-Aug; fall, Sep-Nov)

Additional characteristics will be defined during the 1-year pre-index baseline period:

- Previous COPD treatments
  - ➤ LAMA monotherapy
  - ► LABA monotherapy
  - ➤ ICS monotherapy
  - ➤ LAMA/ICS free combination therapy
- Use of other respiratory drugs
  - Mucolytics
  - > Theophylline
  - ➤ Short-acting beta-agonists
  - Short-acting muscarinic antagonists
- Previous acute COPD exacerbation (measured both 12 months and in the 30 days prior to cohort entry), categorized as 0, 1, or 2+.
  - ➤ All exacerbations (Moderate+Severe)
  - An outpatient visit with a diagnosis code for COPD in any field + a prescription for an oral corticosteroid or an antibiotic for respiratory infections (Moderate); prescriptions within 30 days of each other were considered as continuation of the initial exacerbation.
  - ► Hospitalizations or emergency room visits with a primary diagnosis for COPD

### Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

(Severe); hospitalizations or emergency room visits within 30 days of each other were considered as continuation of the initial exacerbation.

- Hospitalizations caused by exacerbation of heart failure in 12 months prior to index date, categorized as
  - **>** 0;
  - **>** 1;
  - **>** 2+.
- All-cause hospitalizations in 12 months prior to index date;
  - ▶ 0;
  - **>** 1;
  - **>** 2+.
- Comorbidities:
  - > Cardiovascular disease
  - Cerebrovascular disease
  - Diabetes
  - Chronic kidney disease
  - Pneumonia
  - Cancer
  - Cirrhosis
- Charlson Comorbidity Index (CCI)
- History of medications dispensed in the 12 months before or on the index date will be identified from the pharmacy dispensing history:
  - > Cardiovascular drugs:

antihypertensives;

antiarrhythmics;

nitrates;

heart failure medications

- > Lipid-lowering medications
- ➤ Blood glucose-lowering medications
- > Anticoagulants and antiplatelet agents
- Antibiotics
- > Antineoplastic agents
- COPD severity

The definition of the severity of COPD in this study was developed based on the information in previous studies, GOLD recommendations and clinical practice in Taiwan, see below. Patients who fulfil criteria for more than one category will be classified as being in the most severe category.

Operational definition of COPD severity:

➤ Mild:

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Naïve to COPD treatment, or at least one dispensing of the following categories of medications either alone or in combination: 1) SABA or SAMA or SABA+SAMA, 2) LAMA or LABA monotherapy, 3) theophylline or mucolytics, in the 12 months before the index date;

#### ➤ Moderate:

At least one dispensing of LAMA + LABA in the 12 months before the index date;

#### > Severe:

Occurrence of at least one of the following events in the 12 months before the index date:

- Hospitalization with a primary diagnosis for COPD
- Hospitalization with a primary diagnosis for pneumonia
- Second course of antibiotics for respiratory tract infections; a single course of antibiotic treatment involving multiple dispensings is defined as that involving consecutive dispensings of antibiotics with fewer than 7 days between the end of days of supply of one dispensing and the date of the next dispensing
- Second course of systemic corticosteroids for the treatment of COPD exacerbation; a single course of systemic corticosteroids involving multiple dispensings is defined as that involving consecutive dispensings with fewer than 7 days between the end of days of supply of one dispensing and the date of the next dispensing.
- Two diagnoses of COPD exacerbation (ICD-10: J44.1; ICD-9: 491.21) without hospitalisation

#### ➤ Very severe:

Occurrence of at least one of the following events in the 12 months before the index date unless other time period is specified:

- Dispensed oxygen therapy
- Dispensed nebuliser therapy

Diagnosis codes and drug codes are listed in the annex.

#### 8. DATA SOURCES

Data sources include Taiwan National Health Insurance (NHI), Taiwan Cancer Registry (TCR) and Taiwan Mortality Data. Taiwan Department of Statistics, Ministry of Health and Welfare is the unit designated by the government to manage health and social welfare statistical databases, and to develop data platform for academic research. Through the services provided by the Health and Welfare Data Science Center (HWDSC) of the Department of Statistics, researchers may access a wide range of health and welfare data, including claims, mortality (with cause of death) and Taiwan Cancer Registry (TCR). The HWDSC staff encrypt the national ID for all individuals according to a secure encryption

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

algorithm that is not made known to the public. The encrypted ID is unique for all individuals and will be used for linkage between databases.

#### 9. DATA MANAGEMENT AND SOFTWARE/TOOLS

#### 9.1 **SOFTWARE/TOOLS**

All analysis will be conducted by Taiwanese collaborators using SAS software version 9.4 (SAS Institute, Inc., Cary, NC).

#### 9.2 HANDLING OF MISSING VALUES

As administrative data routinely submitted to the health authority, there are no missing value in the health insurance claims. Handling of apparently inconsistent is described under section 9.3. The small number of subjects with missing information on date of birth or gender will be excluded from the study and described in Figure 1.

#### 9.3 HANDLING OF INCONSISTENCIES IN DATA AND OUTLIERS

No clinical parameter values (such as blood pressure or laboratory examination results) are available, therefore potential outliers of continuous variables are not a major concern. Apparently inconsistent data, such birth year of 1860 or Tio+Olo prescriptions during the years that it was not covered, would be identified and subjects with inconsistent data will be excluded from analysis and described in <u>Figure 1</u>.

#### 10. DATA ANALYSIS

#### 10.1 MAIN ANALYSIS

All variables, including patient characteristics, baseline measures, and outcomes, will be analyzed descriptively.

• For all analyses, variables will be reported as follows: Continuous variables (e.g., age) will be presented as means (with standard deviation, SD) and/or medians (with interquartile range, IQR), minimum, maximum.

### Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

• Categorical variables (e.g., sex) will be presented as absolute and relative frequencies.

All analyses will be presented for each treatment group (Tio+Olo vs LABA/ICS) overall. We will first describe formation of the study cohort. Propensity score (PS) matching will be used to generate two comparable treatment groups. All covariates, except season of index date, will be used to estimate the propensity score with logistic regression. Patients in LABA/ICS group will be individually matched to patients in the Tio/Olo group with 1:1 ratio. A caliper of 0.06 standard deviation of logit (propensity score) will be used to define the range of estimated PS within which to select the comparator. Within that range the LABA/ICS patient with the closest estimated propensity score to the Tio/Olo patient will be selected.

Patient characteristics at baseline in patients treated with Tio+Olo and patients treated with LABA/ICS will be described separately using standard descriptive statistics after propensity score matching. Absolute standardized differences (ASDs) will be used to compare the characteristics between the two groups after propensity score matching, in which a >0.1 ASD indicates a meaningful difference.

All the analyses for primary outcome and secondary outcomes will be performed on patients after propensity score matching. Baseline characteristic table shell are provided in <u>Table 1</u>. The propensity score matching will be carried out once without re-matching.

For the analysis of the primary outcome, individuals will be followed up from the index date until the first moderate or severe COPD exacerbation. The data after the earliest date of the following event would be censored:

- 1) disenrollment
- 2) the end of the study period
- 3) death
- 4) discontinuation of index drug use (a lapse of 45 days without subsequent prescription)
- 5) switching from Tio/Olo to ICS/LABA or from ICS/LABA to Tio/Olo
- 6) escalation to triple therapies (ICS/LAMA/LABA free or fix dose combination) Note that per study protocol, switching from one ICS/LABA to another ICS/LABA is not a censoring event.

Univariate proportional hazard regression model will be used to compare the time to event between the two treatment groups. It will provide an estimate of the hazard ratio (HR) of time to the first moderate or severe COPD exacerbation associated with Tio+Olo use relative to LABA/ICS use, along with 95% CI. In the event that there are baseline covariates with unequal distribution between the treatment groups, defined as absolute standardized difference larger than 0.1, the covariate(s) will be included in a multiple regression model in addition to the exposure status (Tio/Olo or LABA/ICS).

The analysis of the secondary objectives related to time to triple therapy escalation and time to first hospitalization for community-acquired pneumonia will be univariate proportional hazard regression model with an as-treated approach, similar to that of the primary analysis. The estimate of hazard ratio (HR) of time to triple therapy escalation and first hospitalization for community-acquired pneumonia associated with Tio+Olo use relative to LABA/ICS use,

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

along with 95% CI will be provided. For the analysis of these time-to-event outcomes, patients will be followed until the event of interest or earliest of the date of the follows, whichever happened first:

- 1) outcome event of interest;
- 2) disenrollment;
- 3) the end of the study period;
- 4) death;
- 5) discontinuation of index drug use (a lapse of 45 days without subsequent prescription)
- 6) switching from Tio/Olo to ICS/LABA or from ICS/LABA to Tio/Olo

In the event that there are baseline covariates with unequal distribution between the treatment groups, defined as absolute standardized difference larger than 0.1, the covariate(s) will be included in a multiple regression model in addition to the exposure status (Tio/Olo or LABA/ICS).

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 



Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The analysis of the secondary objectives related to annualized rate of prescriptions of rescue medications, the rate ratio of Tio+Olo – exposed group relative to LABA/ICS group, along with 95% CIs will be derived using univariate negative binomial model. Individuals in the study cohort will be followed from the index date until the earliest of the date of:

- 1) disenrollment;
- 2) the end of the study period;
- 3) death;
- 4) discontinuation of the index drug use (a lapse of 45 days without subsequent prescription);
- 5) switching from Tio/Olo to ICS/LABA or from ICS/LABA to Tio/Olo

In the event that there are baseline covariates with unequal distribution between the treatment groups, defined as absolute standardized difference larger than 0.1, the covariate(s) will be included in a multiple regression model in addition to the exposure status (Tio/Olo or LABA/ICS).

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



For incidence rates, it will be calculated for each cohort as follows: Incidence rate among the Tio+Olo cohort = (total number of patients in the Tio+Olo cohort experiencing an event of interest for the first time during the given time period) / (total person-time at risk from current use of Tio+Olo during the given period)

### Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Incidence rate among the comparison cohort = (total number of patients in the comparator LABA/ICS cohort experiencing an event of interest for the first time during the given time period) / (total person-time at risk from current use of comparator LABA/ICS during the given period)

The incidence rate ratio (IRR) and incidence difference for the outcome in the Tio+Olo - exposed group relative to that in the comparator group will be derived as follows:

Incidence rate ratio = incidence rate from the Tio+Olo cohort divided by the incidence rate from the matched comparator cohort.

Incidence difference = incidence rate from the Tio+Olo cohort – incidence rate from the matched comparator cohort

For annualized rates, it will be calculated for each cohort as follows: Annualized rate among the Tio+Olo cohort = (total number of events in the Tio+Olo cohort during the given time period) / (total person-year at risk from current use of Tio+Olo during the given period)

Annualized rate among the comparison cohort = (total number of events in the comparator LABA/ICS cohort during the given time period) / (total person-year at risk from current use of comparator LABA/ICS during the given period)

The incidence rate ratio (IRR) for the triple therapy initiation in the Tio+Olo - exposed group relative to that in the comparator group, along with 95% CIs will be derived using univariate negative binomial model. In the event that there are baseline covariates with unequal distribution between the treatment groups, defined as absolute standardized difference larger than 0.1, the covariate(s) will be included in a multiple regression model in addition to the exposure status (Tio/Olo or LABA/ICS).

For annualized rate of moderate or severe COPD exacerbations and annualized rate of prescriptions of rescue medications, the ratio of Tio+Olo – exposed group relative to LABA/ICS group, along with 95% CIs will be derived using negative binomial model. In the event that there are baseline covariates with unequal distribution between the treatment groups, defined as absolute standardized difference larger than 0.1, the covariate(s) will be included in a multiple regression model in addition to the exposure status (Tio/Olo or LABA/ICS).

SAS codes for negative binominal model are provided in Annex.



Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



#### 10.3 SAFETY ANALYSIS

Not applicable.

## 11. QUALITY CONTROL

Greater details are documented in the NIS-DMRP.

### 12. REFERENCES

#### 12.1 PUBLISHED REFERENCES

- **P21-01394** Global initiative for chronic obstructive lung disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease (2021 REPORT) . https://goldcopd.org/goldreports/.
- **P07-11820** Wedzicha JA et al. The prevention of COPD exacerbations by salmeterol/fluticasone propionate or tiotropium bromide. Am J Respir Crit Care Med.2008;177:19-26.
- **P16-05628** Wedzicha J A, et al. Indacaterol–Glycopyrronium versus Salmeterol–Fluticasone for COPD. N Engl J Med, 2016, 2016(374): 2222-2234

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 12.2 UNPUBLISHED REFERENCES

None

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### ANNEX 1. ADDITIONAL INFORMATION

Table 1. Baseline characteristic of the study cohort

| | Before propensity score match | | | natch | After propensity score mate | | | natch | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Tio | /Olo | ICS/I | LABA | | Tio | /Olo | ICS/L | ABA | |
| | coł | ort | coł | nort | ASD | coh | ort | coh | ort | ASD |
| | N | % | N | % | | N | % | N | % | 1Mo |
| Gender | | | | | | | | | | |
| Male | | | | | | | | | | |
| Female | | | | | | | | | | |
| Age | | | | | | | | | | |
| 40~54 | | | | | | | | | | |
| 55~69 | | | | | | | | | | |
| 70~84 | | | | | | | | | | |
| 85+ | | | | | | | | | | |
| Calendar year of cohort entry | | | | | | | | | | |
| 2014 | | | | | | | | | | |
| 2015 | | | | | | | | | | |
| 2016 | | | | | | | | | | |
| 2017 | | | | | | | | | | |
| 2018 | | | | | | | | | | |
| 2019 | | | | | | | | | | |
| Season of index date | | | | | | | | | | |
| Spring (Mar-May) | | | | | | | | | | |
| Summer (Jun-Aug) | | | | | | | | | | |
| Fall (Sep-Nov) | | | | | | | | | | |
| Winter (Dec-Feb) | | | | | | | | | | |
| COPD treatments in 1 year prior | | | | | | | | | | |
| to index date | | | | | | | | | | |
| LAMA | | | | | | | | | | |
| LABA | | | | | | | | | | |
| ICS | | | | | | | | | | |
| ICS+LAMA free combination | | | | | | | | | | |
| Use of other respiratory drugs in | 1 year | prior | | | | | | | | |
| to index date | | | | | | | | | | |
| Mucolytics | | | | | | | | | | |
| Theophylline | | | | | | | | | | |
| Short-acting beta-agonists | | | | | | | | | | |
| (SABA) | | | | | | | | | | |
| Short-acting muscarinic antagonists (SAMA) | | | | | | | | | | |
| antagonists (SAIVIA) | | | | | | | | | | |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

| | Before propensity score match | | | After propensity score match | | |
|---|---|---|---|---|---|---|
| | Tio/Olo | ICS/LABA | | Tio/Olo | ICS/LABA | |
| | cohort | cohort | ASD | cohort | cohort | ASD |
| | N % | N % | | N % | N % | |
| Acute COPD exacerbation in 1 years | ear prior to | | | | | |
| index date | | | | | | |
| Moderate exacerbation | | | | | | |
| 0 | | | | | | |
| 1 | | | | | | |
| >=2 | | | | | | |
| Severe exacerbation | | | | | | |
| 0 | | | | | | |
| 1 | | | | | | |
| >=2 | | | | | | |
| All exacerbations (Moderate | | | | | | |
| + Severe) | | | | | | |
| 0 | | | | | | |
| 1 | | | | | | |
| >=2 | | | | | | |
| Acute COPD exacerbation in the | 30 days prior | | | | | |
| to index date | | | | | | |
| Moderate exacerbation | | | | | | |
| 0 | | | | | | |
| 1 | | | | | | |
| >=2 | | | | | | |
| Severe exacerbation | | | | | | |
| 0 | | | | | | |
| 1 | | | | | | |
| >=2 | | | | | | |
| All exacerbations (Moderate | | | | | | |
| + Severe) | | | | | | |
| 0 | | | | | | |
| 1 | | | | | | |
| >=2 | | | | | | |
| Hospitalizations caused by exact index date | erbation of COI | PD in 1 year p | rior to | | | |
| 0 | | | | | | |
| 1 | | | | | | |
| >=2 | or prior to | | | | | |
| All-cause hospitalizations in 1 ye<br>index date | ear prior to | | | | | |
| 0 | | | | | | |
| ~ | | | | | | |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

| | Before propensity score match | | | After propensity score ma | | | natch | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Tio | Tio/Olo<br>cohort | | LABA | | Tio | /Olo | ICS/I | ABA | |
| | col | | | nort | ASD | cohort | | cohort | | ASD |
| | N | % | N | % | | N | % | N | % | |
| 1 | | | | | | | | | | |
| >=2 | | | | | | | | | | |
| Comorbidities: | | | | | | | | | | |
| Cardiovascular disease | | | | | | | | | | |
| Cerebrovascular disease | | | | | | | | | | |
| Diabetes | | | | | | | | | | |
| Chronic kidney disease | | | | | | | | | | |
| Pneumonia | | | | | | | | | | |
| Cancer | | | | | | | | | | |
| Cirrhosis | | | | | | | | | | |
| Charlson Comorbidity Index (CCI) | | | | | | | | | | |
| History of medications dispensed | d in 1 ye | ar prio | r to inc | dex | | | | | | |
| date | | | | | | | | | | |
| Cardiovascular drugs: | | | | | | | | | | |
| Antihypertensives | | | | | | | | | | |
| Antiarrhythmics | | | | | | | | | | |
| Nitrates | | | | | | | | | | |
| Heart failure medications | | | | | | | | | | |
| Lipid-lowering medications | | | | | | | | | | |
| Blood glucose-lowering | | | | | | | | | | |
| medications | | | | | | | | | | |
| Anticoagulants and antiplatelet agents | | | | | | | | | | |
| Antibiotics | | | | | | | | | | |
| Antineoplastic agents | | | | | | | | | | |
| COPD severity | | | | | | | | | | |
| Mild | | | | | | | | | | |
| Moderate | | | | | | | | | | |
| Severe | | | | | | | | | | |
| Very severe | | | | | | | | | | |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Table 2. Hazard ratios for COPD exacerbation, Tio/Olo users vs. ICS/LABA users

| After PS match | Moderate exacerbation | Severe exacerbation | All exacerbation<br>(Moderate + Severe) |
|---|---|---|---|
| | HR (95% CI) | HR (95% CI) | HR (95% CI) |
| Tio/Olo | | | |
| ICS/LABA | Reference | Reference | Reference |
| | Adjusted* HR (95% CI) | Adjusted* HR (95% CI) | Adjusted* HR (95% CI) |
| Tio/Olo | Adjusted* HR (95% CI) | Adjusted* HR (95% CI) | Adjusted* HR (95% CI) |

<sup>\*</sup> If needed, list of adjusted covariates will be listed.

Table 3. Hazard ratio for time to first triple therapy escalation, Tio/Olo users vs. ICS/LABA users

| A 64 DC + - - | Triple the | rapy escalation |
|----------------|-------------|-----------------------|
| After PS match | HR (95% CI) | Adjusted* HR (95% CI) |
| Tio/Olo | | |
| ICS/LABA | Reference | Reference |

<sup>\*</sup> If needed, list of adjusted covariates will be listed.

Table 4. Incidence rates of triple therapy initiation among the two cohorts, incidence rate ratio and incidence difference estimates

| After PS match | No.<br>with<br>events | Person-<br>years | Incidence<br>Rate<br>(95% CI) | IRR<br>(95% CI) | Adjusted*<br>IRR<br>(95% CI) | Incidence<br>difference<br>(95% CI) |
|---|---|---|---|---|---|---|
| Triple therapy escalation | | | | | | |
| Tio/Olo | | | | | | |
| ICS/LABA | | | | Reference | Reference | Reference |

<sup>\*</sup> If needed, list of adjusted covariates will be listed.

Table 5. Hazard ratio for time to first hospitalization for community-acquired pneumonia, Tio/Olo users vs. ICS/LABA users

| After PS match | Hospitalization for community-acquired pneumonia | |
|---|---|---|
| After P5 match | HR (95% CI) | Adjusted* HR (95% CI) |
| Tio/Olo | | |
| ICS/LABA | Reference | Reference |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Table 6. Annualized rates of prescription of rescue medications and moderate or severe COPD exacerbations

| After PS match | No. of<br>patients<br>with<br>events | No. of events | Person-<br>years | Annualized<br>rate<br>(95CI) | Annualized<br>rate ratio<br>(95CI) | Adjusted*<br>rate ratio<br>(95CI) |
|---|---|---|---|---|---|---|
| Rescue medication | | | | | | |
| Tio/Olo | | | | | | |
| ICS/LABA | | | | | Reference | Reference |
| Moderate exacerbation | | | | | | |
| Tio/Olo | | | | | | |
| ICS/LABA | | | | | Reference | Reference |
| Severe exacerbation | | | | | | |
| Tio/Olo | | | | | | |
| ICS/LABA | | | | | Reference | Reference |
| All exacerbation | | | | | | |
| (Moderate + Severe) | | | | | | |
| Tio/Olo | | | | | | |
| ICS/LABA | | | | | Reference | Reference |

<sup>\*</sup> If needed, list of adjusted covariates will be listed.

<sup>\*</sup> If needed, list of adjusted covariates will be listed.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Appendix 1. SAS code template for negative binominal model in the analysis of the secondary outcomes of interest

The following codes are provided by Boehringer Ingelheim statistician

PROC GENMOD DATA=test; CLASS treat (ref='LABA/ICS') cova\_cat; MODEL ep\_count = treat cova\_cat cova\_con / DIST=negbin LINK=LOGTYPE3 OFFSET=logt; LSMEANS treat / DIFF CL; ESTIMATE 'Treatment effect on ratio-scale' treat 1 -1 / EXP; RUN;

(In the model,

treat: Tio+Olo group OR LABA/ICS group;

Cova\_cat: categorical covariates; Cova\_con: continuous covariates)

For univariate analysis, Cova cat and Cova con are not applicable.

For calculating incidence rate ratio with 95% CI of triple therapy initiation (Tio+Olo vs. LABA/ICS),

ep\_count (response): 1 (triple therapy initiation occurred per patient) or 0 (triple therapy initiation not occurred per patient);

logt: nature log of the time at risk (first event per patient)

For calculating ratio (with 95% CI) of annualized rate of moderate or severe COPD exacerbations and annualized rate of prescriptions of rescue medications (Tio+Olo vs. LABA/ICS),

ep\_count (response): number of events per patient logt: nature log of the time at risk per patient

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Appendix 2. ICD-9/10-CM codes and procedure codes for identification of study cohorts

| | ICD9 | ICD10 |
|---|---|---|
| For inclusion criteria | | |
| COPD | 491.x, 492.x, 496 | J41.x, J42, J43.x, J44.x |
| For exclusion criteria | | |
| Asthma | 493.x | J45.x |
| Allergic rhinitis | 477.x | J30.x |
| Lung cancer | 162.x | C33.x, C34.x, C7A.090, |
| | | D02.2 |
| Interstitial lung disease | 238.1, 500, 501, 502, 503, | J60, J61, J62.x, J63.x, J64, |
| | 504, 505, 506.4, 508.1, | J65, J66.x, J68.4, J70.x (no |
| | 508.8, 515, 516.x | 70.2), J84.1x (no J84.114), |
| | | J84.2, J84.3, J84.89, J84.9, |
| | | J94.1 |

| <b>Procedure codes</b> | Content |
|---|---|
| 68037A | Lung transplantation |
| 68037B | Lung transplantation - Unilateral lung |
| 68047B | Lung transplantation - bilateral sequential or en bloc double lung |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## Appendix 3. COPD medications

| Groups | Drug name | ATC code |
|---|---|---|
| LAMA | Tiotropium bromide | R03BB04 |
| | Glycopyrrolate | R03BB06 |
| | Umeclidinium | R03BB07 |
| LABA | Salmeterol | R03AC12 |
| | Formoterol | R03AC13 |
| | Procaterol | R03AC16 |
| | Indacaterol | R03AC18 |
| | Olodaterol | R03AC19 |
| ICS | Beclometasone(=beclomethasone) | R03BA01 |
| | Budesonide | R03BA02 |
| | Fluticasone | R03BA05 |
| | Ciclesonide | R03BA08 |
| ICS/LABA | Salmeterol and Fluticasone | R03AK06 |
| | Formoterol and Budesonide | R03AK07 |
| | Formoterol and Beclometasone | R03AK08 |
| | Vilanterol and Fluticasone furoate | R03AK10 |
| | Formoterol and Fluticasone | R03AK11 |
| LABA/LAMA | Vilanterol and Umeclidinium<br>bromide | R03AL03 |
| | Indacaterol and Glycopyrronium | R03AL04 |
| | bromide<br>Olodaterol and Tiotropium | R03AL06 |
| 8 | bromide | |
| LABA/LAMA/ICS | Vilanterol, Umeclidinium bromide<br>and Fluticasone furoate | R03AL08 |
| | Formoterol, Glycopyrronium | R03AL09 |
| | bromide and Beclometasone | |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## Appendix 4. ICD codes and operational definition of comorbidities

| | Comorbidities: | ICD codes | Operational definition |
|---|---|---|---|
| 1. | Diabetes | ICD9: 250 | Either inpatient diagnosis or |
| | | ICD10: E10.x-E11.x | more than twice outpatient |
| | | | diagnosis |
| 2. | Cardiovascular disease | ICD9: 250.7, 401-405, | Either inpatient diagnosis or |
| | | 410-414, 425-428, 429.1- | more than twice outpatient |
| | | 429.3, 441, 442, 458 | diagnosis |
| | | ICD10: E10.5x, E11.5x, | |
| | | 110- 13.x, 15.x, 20.x- | |
| | | 122.x, 124.x, 125.x, 142.x- | |
| | | 144, 145.xx, 146.x-149.x, | |
| | | I50.xx, I51.5, I51.7, I51.9, | |
| | | 171.xx, 179.0, 172.x, | |
| | | 177.7x, 195.x | |
| 3. | Cerebrovascular disease | ICD9: 430-438 | Either inpatient diagnosis or |
| | | ICD10: 160.x-163.x, 165.x, | more than twice outpatient |
| | | 166.x, G45.x, G46.x, 167.x- | diagnosis |
| | | 169.x | |
| 4. | Cancer | ICD9: 140-199, 200-208 | Inpatient diagnosis. |
| | | ICD10: C00-C26, C30-34, | |
| | | C37-39, C40-41, C43-49, | |
| | | C4A, C50-58, C60-69, | |
| | | C70-79,C7A, C7B, C80- | |
| | | 86, C88, C90-96, | |
| 5. | Chronic kidney disease | ICD9: 585-587, | Either inpatient diagnosis or |
| | | ICD10: N18-19, N26.1, | more than twice outpatient |
| | | N26.9 | diagnosis |
| 6. | Pneumonia | ICD9: 480-486, 487.0 | Inpatient diagnosis |
| | | ICD10: J10.0, J11.0, J12- | |
| <u></u> | | J18, | |
| 7. | Cirrhosis | | Either inpatient diagnosis or |
| | | ICD10: K70.3x, K74.3, | more than twice outpatient |
| | | K74.4, K74.5, K74.6x | diagnosis |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## Appendix 5. Drugs of interest

| Groups | ATC code |
|---|---|
| Use of other respirato | Use of other respiratory drugs |
| Mucolytics | R05CB, R05CB01, R05CB02, R05CB03, R05CB04, R05CB05, |
| | R05CB06, R05CB10, R05CB11, R05CB91, R05CB92 |
| Theophylline | R03DA04, R03DA54, R03DA74, R03DB04 |
| SABA | R03AC02, R03AC03, R03AC04, R03AC06 |
| SAMA | R03BB01 |
| SABA/SAMA | R03AL01, R03AL02 |
| Drugs for COPD exac | erbation treatment |
| Oral corticosteroid | H02AB01, H02AB02, H02AB04, H02AB05, H02AB06, H02AB08, |
| | H02AB10, H02BX, H02BX91 |
| Antibiotic for COPD | J01AA02, J01CA04, J01CR02, J01CR05, J01EE01, J01DC01, |
| exacerbation | J01DC02, J01DC03, J01DC04, J01DC05, J01DC06, J01DC07, |
| | J01DC09, J01DC14, J01DD01, J01DD02, J01DD04, J01DD05, |
| | J01DD06, J01DD07, J01DD08, J01DD12, J01DD13, J01DD14, |
| | J01DD52, J01DD62, J01DE01, J01DE02, J01FA01, J01EA02, |
| | J01EA03, J01EA06, J01EA07, J01EA08, J01FA09, J01FA10, |
| | J01FA15, J01FA91, J01MA01, J01MA02, J01MA03, J01MA04, |
| | J01MA06, J01MA07, J01MA09, J01MA12, J01MA14, J01MA15 |
| Drugs for Medication history | |
| <ul> <li>Cardiovascular d</li> </ul> | rugs |
| Anti-hypertensives | C02AA01, C02AA02, C02AA04, C02AB01, C02AB02, C02AC01, |
| | C02CA01, C02CA04, C02CA, C02CC02, C02DA01, C02DB02, |
| | C02DC01, C02DD01, C02LA01, C02LA50, C02LA51, C02LB01, |
| | C02LG02, C02N, C03AA01, C03AA03, C03AA06, C03AA07, |
| | C03AA, C03BA04, C03BA08, C03BA11, C03CA01, C03CA02, |
| | C03CA04, C03CC01, C03DA01, C03DA04, C03DB01, C03DB02, |
| | C03EA01, C03EA, C07AA01, C07AA02, C07AA03, C07AA05, |
| | C07AA06, C07AA07, C07AA12, C07AA15, C07AA19, C07AB02, |
| | C07AB03, C07AB04, C07AB05, C07AB07, C07AB09, C07AB12, |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

| | C10AX13, C10AX14, C10AX |
|---|---|
| | C10AD02, C10AD03, C10AD06, C10AD, C10AX02, C10AX09, |
| | C10AB06, C10AB09, C10AC01, C10AC02, C10AC03, C10AD01, |
| Agents, Plain | C10AA08, C10AB01, C10AB02, C10AB03, C10AB04, C10AB05, |
| Lipid Modifying | C10AA01, C10AA02, C10AA03, C10AA04, C10AA05, C10AA07, |
| <ul><li>Lipid-lowering</li></ul> | medications |
| Nitrates | C01DA02, C01DA05, C01DA08, C01DA14 |
| | C09CA07, C09CA08, C09CA09 |
| | C09AA16, C09CA01, C09CA02, C09CA03, C09CA04, C09CA06, |
| | C09AA04, C09AA05, C09AA06, C09AA07, C09AA08, C09AA09, |
| | C03CA04, C03DA04, C07AG02, C09AA01, C09AA02, C09AA03, |
| medications | C01CA02, C01CA07, C01CE02, C01EB09, C01EB17, C03CA02, |
| Heart failure | C01AA04, C01AA05, C01AA07, C01AA08, C01AB01, C01AC01, |
| | C07AB12, C08DA01, C08DB01 |
| | C07AB02, C07AB03, C07AB04, C07AB05, C07AB07, C07AB09, |
| | C07AA03, C07AA05, C07AA07, C07AA12, C07AA15, C07AA19, |
| | C01CA04, C01CA06, C01EB10, C01EB17, C07AA01, C07AA02, |
| | C01BB02, C01BC03, C01BC04, C01BD01, C01BD07, C01CA02, |
| | C01BA01, C01BA02, C01BA03, C01BA04, C01BA08, C01BB01, |
| Antiarrhythmics | C01AA04, C01AA05, C01AA07, C01AA08, C01AB01, C01AC01, |
| | C09XA52, C09XA53, C09XA54 |
| | C09DB04, C09DB07, C09DX01, C09DX03, C09DX04, C09XA02, |
| | C09DA06, C09DA07, C09DA08, C09DA09, C09DB01, C09DB02 |
| | C09CA07, C09CA08, C09CA09, C09DA01, C09DA03, C09DA04 |
| | C09BB, C09CA01, C09CA02, C09CA03, C09CA04, C09CA06 |
| | C09BA01, C09BA02, C09BA04, C09BB04, C09BB05, C09BB |
| | C09AA05, C09AA06, C09AA07, C09AA08, C09AA09, C09AA16. |
| | C08DA01, C08DB01, C09AA01, C09AA02, C09AA03, C09AA04. |
| | C08CA07, C08CA08, C08CA09, C08CA12, C08CA13, C08CA15 |
| | C07DA06, C08CA01, C08CA02, C08CA03, C08CA04, C08CA05 |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

| Lipid Modifying | C10BA01, C10BA02, C10BA03, C10BA05, C10BX03 |
|---|---|
| Agents, Combinations | |
| Blood glucose-low | ering medications |
| Insulins and analogues | A10AB01, A10AB03, A10AB04, A10AB05, A10AB06, A10AB30, |
| | A10AC01, A10AC03, A10AC30, A10AD01, A10AD03, |
| | A10AD04, A10AD05, A10AD06, A10AE01, A10AE04, A10AE05, |
| | A10AE06, A10AE54 |
| ٥ | A10BA02, A10BA03, A10BB01, A10BB02, A10BB03, A10BB04, |
| drugs, excl. insulins | A10BB05, A10BB07, A10BB08, A10BB09, A10BB12, A10BB31, |
| | A10BD02, A10BD03, A10BD05, A10BD07, A10BD08, A10BD09, |
| | A10BD10, A10BD11, A10BD13, A10BD14, A10BD, A10BD15, |
| | A10BD19, A10BD20, A10BD21, A10BD24, A10BF01, A10BF02, |
| | A10BG02, A10BG03, A10BH01, A10BH02, A10BH03, A10BH04, |
| | A10BH05, A10BJ01, A10BJ02, A10BJ03, A10BJ05, A10BJ06, |
| | A10BK01, A10BK02, A10BK03, A10BK04, A10BX01, A10BX02, |
| | A10BX03, A10BX08 |
| <ul> <li>Anticoagulants an</li> </ul> | d antiplatelet agents |
| Vitamin K antagonists | B01AA02, B01AA03 |
| Heparin group | B01AB01, B01AB04, B01AB05, B01AB06, B01AB10 |
| Platelet aggregation | B01AC04, B01AC05, B01AC06, B01AC07, B01AC09, B01AC11, |
| inhibitors excl. heparin | B01AC13, B01AC16, B01AC17, B01AC21, B01AC22, B01AC23, |
| | B01AC24, B01AC27, B01AC30 |
| Enzymes | B01AD01, B01AD02, B01AD04, B01AD10, B01AD11 |
| Direct thrombin | B01AE07 |
| inhibitors | |
| Direct factor Xa | B01AF01, B01AF02, B01AF03 |
| inhibitors | |
| Other antithrombotic | B01AX05 |
| agents | |
| <ul> <li>Antibiotic</li> </ul> | 1 |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

| Antibacterials for | J01AA01, J01AA02, J01AA03, J01AA04, J01AA06, J01AA07, |
|---|---|
| systemic use | J01AA08, J01AA09, J01AA12, J01AA56, J01BA01, J01BA02, |
| | J01BA51, J01CA01, J01CA02, J01CA03, J01CA04, J01CA06, |
| | J01CA08, J01CA09, J01CA10, J01CA12, J01CA13, J01CA14, |
| | J01CA15, J01CA16, J01CA18, J01CA20, J01CA91, J01CE01, |
| | J01CE02, J01CE08, J01CE09, J01CE30, J01CF01, J01CF02, |
| | J01CF04, J01CF05, J01CG01, J01CR01, J01CR02, J01CR03, |
| | J01CR04, J01CR05, J01CR50, J01CR50, J01CR50, J01DB01, |
| | J01DB02, J01DB03, J01DB04, J01DB05, J01DB06, J01DB07, |
| | J01DB08, J01DB09, J01DC01, J01DC02, J01DC03, J01DC04, |
| | J01DC05, J01DC06, J01DC07, J01DC09, J01DC14, J01DD01, |
| | J01DD02, J01DD04, J01DD05, J01DD06, J01DD07, J01DD08, |
| | J01DD12, J01DD13, J01DD14, J01DD52, J01DD62, J01DE01, |
| | J01DE02, J01DF01, J01DH02, J01DH03, J01DH04, J01DH51, |
| | J01DI02, J01DI54, J01E, J01EA01, J01EB01, J01EB02, J01EB05, |
| | J01EB06, J01EB20, J01EC, J01EC01, J01EC02, J01EC20, |
| | J01ED01, J01ED05, J01ED20, J01EE01, J01FA01, J01EA02, |
| | J01EA03, J01EA06, J01EA07, J01EA08, J01FA09, J01FA10, |
| | J01FA15, J01FA91, J01FF01, J01FF02, J01GA01, J01GB01, |
| | J01GB03, J01GB04, J01GB05, J01GB06, J01GB07, J01GB08, |
| | J01GB09, J01GB11, J01MA01, J01MA02, J01MA03, J01MA04, |
| | J01MA06, J01MA07, J01MA09, J01MA12, J01MA14, J01MA15, |
| | J01MB01, J01MB02, J01MB03, J01MB04, J01MB08, J01RA02, |
| | J01XA01, J01XA02, J01XB, J01XB01, J01XC01, J01XD01, |
| | J01XD02, J01XD03, J01XE, J01XE01, J01XE02, J01XX01, |
| | J01XX04, J01XX05, J01XX07, J01XX08, J01XX09, J01XX91 |
| Antimycotics for | J02AA01, J02AB01, J02AB02, J02AC01, J02AC02, J02AC03, |
| systemic use | J02AC04, J02AC05, J02AX01, J02AX04, J02AX05, J02AX06 |
| Antimycobacterials | J04AA03, J04AB01, J04AB02, J04AB03, J04AB04, J04AB91, |
| | J04AC01, J04AC51, J04AD01, J04AK01, J04AK02, J04AK04, |
| | J04AM02, J04AM03, J04AM05, J04AM06, J04AM07, J04BA01, |
| | J04BA02 |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

| Antineoplastic age | ents |
|---|---|
| Alkylating agents | L01AA01, L01AA02, L01AA03, L01AA06, L01AA09, L01AB01, |
| | L01AC01, L01AC03, L01AD01, L01AD02, L01AD06, L01AX03, |
| | L01AX04 |
| Antimetabolites | L01BA01, L01BA04, L01BA05, L01BB02, L01BB03, L01BB04, |
| | L01BB05, L01BB06, L01BC01, L01BC02, L01BC03, L01BC05, |
| | L01BC06, L01BC07, L01BC53, L01BC59 |
| Plant alkaloids and | L01CA01,L01CA02, L01CA04, L01CB01, L01CD01, L01CD02, |
| other natural products | L01CE01, L01CE02 |
| Cytotoxic antibiotics | L01DA01, L01DB01, L01DB02, L01DB03, L01DB04, L01DB06, |
| and related substances | L01DB07, L01DC01, L01DC03, L01DC04 |
| Protein kinase inhibitors | L01EA01, L01EA02, L01EA03, L01EA05, L01EB01, L01EB02, |
| | L01EB03, L01EB04, L01EB07, L01EC01, L01EC02, L01ED01, |
| | L01ED02, L01ED03, L01ED04, L01ED05, L01EE01, L01EF01, |
| | L01EF02, L01EG01, L01EG02, L01EH01, L01EJ01, L01EK01, |
| | L01EL01, L01EM02, L01EX01, L01EX02, L01EX03, L01EX04, |
| | L01EX05, L01EX07, L01EX08, L01EX09, L01EX10, L01EX14 |
| Other antineoplastic | L01XA01, L01XA02, L01XA03, L01XB01, L01XC02, L01XC03, |
| agents | L01XC06, L01XC07, L01XC08, L01XC12, L01XC13, L01XC14, |
| | L01XC15, L01XC17, L01XC18, L01XC19, L01XC21, L01XC24, |
| | L01XC26, L01XC31, L01XC32, L01XF01, L01XG01, L01XG02, |
| | L01XG03, L01XK01, L01XK04, L01XX02, L01XX05, L01XX11, |
| | L01XX23, L01XX27, L01XX35, L01XX41, L01XX52, L01XX |
| Hormones and related | L02AA01, L02AA91, L02AB01, L02AB02, L02AE01, L02AE02, |
| agents | L02AE03, L02AE04 |
| Hormone antagonists | L02BA01, L02BA02, L02BB01, L02BB03, L02BB04, L02BB05, |
| and related agents | L02BG01, L02BG03, L02BG04, L02BG06, L02BX02, L02BX03 |
| | I |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## Appendix 6. Procedure codes for oxygen therapy or nebuliser therapy

| Description | Procedure codes |
|---|---|
| Oxygen therapy | 47054C, 54007C1, 57001B, 57002B, 57003C, 57004C, 57019C, 57020C, 57023B, 57029C |
| Nebuliser therapy | 57021C, 57022C, 57024B |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c40729787-01 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### ANNEX 2. REVIEWERS AND APPROVAL SIGNATURES

The NIS SEAP must be sent for review to the following individuals prior to approval.

| Reviewer | NIS involving BI product(s) | NIS not involving BI product(s) | |
|---|---|---|---|
| | | Global NIS | Local NIS |
| NIS Lead | X | X | X |
| Global TM Epi* | X | X | X |
| NIS Data Manager | X | X | X |
| TSTAT<br>(for NISnd only) | X | X | X |
| RWE CoE | X | X | |

<sup>\*</sup> When BI NIS lead is not TM Epi

Study Title: Effectiveness of Maintenance Treatment with Tiotropium + Olodaterol in Comparison to Inhaled Corticosteroids + Long-acting  $\beta 2$  agonists in COPD patients in Taiwan: a non-interventional study based on the Taiwan National Health Insurance (NHI) data.

**Study Number: 1237-0110** 

Protocol Version: 1.0

I herewith certify that I agree to the content of the study SEAP and to all documents referenced in the study SEAP.

| Position: | Name/Date: | Signature: |
|-----------|------------|------------|
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |